CLINICAL TRIAL: NCT02979483
Title: Management of Symptomatic Advanced Pancreatic Adenocarcinoma: "Urgence Pancreas" - A Prospective A.R.CA.D Cohort Study
Brief Title: Management of Symptomatic Advanced Pancreatic Adenocarcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Urgence Pancreas D16-1
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pancreas; Management Supportive Care Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 14-day emergency integrative supportive care program (14-EISCP) (Experimental): The 14-EISCP starts with the end of visit 1:
  * The investigator must determine which procedures have to be undertaken within the following 14 days (+/- 2 days):
  * Pain management,
  * Nutritional management,
  * Pathological examination and site of biopsy,
  * Imaging,
  * Endoscopy for diagnosis purpose or for biliary/duodenal stenting.
  At the end of the visit the investigator must plan all the supportive care and procedures indicated for the patient and indicate those within a specific form
  Interventions: Other: 14-EISCP

INTERVENTIONS:
Other: 14-EISCP — The 14-EISCP starts with the end of the first visit medical for patients who have symptoms suspicious of or confirmed symptomatic aPDAC (ECOG PS ≥ 2 and/or initially ineligible for clinical trial, FOLFIRINOX or gemcitabine + nab-paclitaxel):
  The The 14-EISCP will include:
  * Pain management,
  * Nutritional management,
  * Pathological examination and site of biopsy,
  * Imaging,
  * Endoscopy for diagnosis purpose or for biliary/duodenal stenting.
  After the 14-EISCP, patients will receive best supportive care or chemotherapy according to their ECOG PS status:
  * ECOG-PS 0-1 and eligible for clinical trial, FOLFIRINOX or gemcitabine + nab-paclitaxel Patient will be treated by : FOLFIRINOX or gemcitabine-nab-paclitaxel or clinical trial
  * ECOG-PS 2-4 and / or ineligible for clinical trial, FOLFIRINOX or gemcitabine + nab-paclitaxel Patients will be treated by: FOLFOX7 lightened

SUMMARY:
This study assessed the feasibility and effects of an early integrative supportive care program in patient with advanced pancreatic adenocarcinoma (aPDAC).

DETAILED DESCRIPTION:
This is a national, multicenter, prospective study, including:

* A 14-day (+/-2 days) integrative supportive care program (14-EISCP) initiated as early as the clinical suspicion of aPDAC,
* Follow-up period after the 14-EISCP.

ECOG PS ≥2 patients with pathologically confirmed or suspected aPDAC on imaging were included at first oncology visit in the 14-EISCP including pain, nutritional, diagnostic and stenting procedures.

Post-EISCP ECOG PS ≤1 patients received mFOLFIRINOX or gemcitabine/nab-paclitaxel, ECOG PS ≥2 patients received mFOLFOX7 or investigator choice chemotherapy or best supportive care.

ELIGIBILITY:
Inclusion criteria

1. Pathologically confirmed or highly suspected aPDAC defined as a pancreatic mass on imaging, suspected distant metastases, no features suggestive of a neuroendocrine tumor, and/or clinico-biological abnormalities compatible with the diagnosis of aPDAC,
2. Age ≥ 18 years,
3. Patients with ECOG PS ≥ 2 and clinico-biological features precluding initial therapeutic clinical trial and/or treatment with FOLFIRINOX or gemcitabine + nab-paclitaxel,
4. No prior history of cancer, except: in situ breast, cervix cancer, or basal cell carcinoma and/or complete remission for more than 3 years from another cancer.
5. Registration in France with the French National Health Care System (CMU included)
6. Patient able to comply with study protocol requirements in the view of the investigator,
7. Before patient registration, written informed consent must be obtained according to ICH/GCP and national/local regulations,
8. Patients requiring at least two components of the integrative care program (pain management, nutritional management, pathological assessment or imaging, and endoscopy/stent).

Exclusion criteria:

1. Any medical, psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial,
2. Patient protected by law,
3. Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-12-19 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
The rate of 14-EISCP success | 14 days (+/- 2 days)
  The success is determined by:
  Program Feasibility :
  The 14-EISCP is considered feasible if the planned procedures, established during the initial consultation with the investigator, is completed within 14 days (+/- 2 days) following the first consultation, or before the start of chemotherapy if it started within 14 days.
  and
  Clinical Benefit at 30 days post-consultation defined by one of the following criteria:
  1. An improvement of ECOG PS from ≥2 to 1 or 0.
  2. A ≥5-point improvement in either fatigue, pain, or global health, as measured by the QLQ-C15-PAL, with no worsening in ECOG PS or the dimensions of fatigue, pain, and global health compared to baseline values.
  3. The initiation of chemotherapy within 30 days of consultation.
  If none of the above criteria (1), (2), or (3) are met, the clinical benefit was considered absent, and the outcome was classified as a failure.
  The success of the 14-EISCP was defined by success of both criteria.

SECONDARY OUTCOMES:
Delay from the first symptom of aPDAC to the first medical appointment | Up to 2-3 months
  Delay between first medical appointment and beginning of chemotherapy in days.
The rate of patients with improved ECOG PS and/or clinico-biological parameters after 14-EISCP. | 14 days; at the end of the 14-EISCP
  The rate of patients with improved ECOG PS and clinico-biologic parameters (liver tests, including bilirubin) at the end of the integrative supportive care program.
The rate of patients receiving chemotherapy and rate of patients with type of chemotherapy effectively given after the 14-EISCP. | At 14 days, at 21 days, up to death
  The rate of patients receiving chemotherapy and rate of patients with type of chemotherapy effectively given after the 14-EISCP.
The mean change of health-related quality of life (HRQoL) score | at 30 days
  The mean change of HRQoL (QLQ-C15-PAL) score between the beginning and the end of the 14-EISCP.
Progression-free survival (PFS) assessment | up to 2 years
  PFS in different patient groups.
Overall survival (OS) assessment | up to 2 years
  OS in different patient groups.
The change of health-related quality of life (HRQoL) | Month 1 and every two months up to two years
  The change of health-related quality of life (HRQoL) as measured by QLQ-C15 PAL. Mean change will be used to compare QoL scores before and after the 14-EISCP.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît ROUSSEAU, MD, Principal Investigator — CHU Henri Mondor Créteil
Locations (12):
- France (12):
  - Institut Sainte Catherine, Avignon
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Léon Bérard, Lyon
  - CH Layne, Mont-de-Marsan
  - Grope Hospitalier Paris Saint Joseph, Paris
  - Hôpital Cochin, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hopitaux du Léman, Thonon-les-Bains
  - CHU Tours - Hôpital Trousseau, Tours